CLINICAL TRIAL: NCT03101774
Title: Effects of Respiratory Physiology-oriented Inspiratory Muscle Training on Respiratory Muscle Function，Quality of Life and Exercise Capacity in Stable COPD With Inspiratory Muscle Weakness: a Randomised Controlled Trial
Brief Title: Inspiratory Muscle Training on Respiratory Muscle Function，Quality of Life and Exercise Capacity in Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weiliang Wu, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuangzhouInsRD
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: COPD
Keywords: inspiratory muscle training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- threshold-IMT group (Experimental): Using inspiratory muscle training using threshold load device for 8 weeks
  Interventions: Device: Threshold inspiratory muscle training
- resisive-IMT group (Experimental): Using inspiratory muscle training using resistive device for 8 weeks
  Interventions: Device: Resistive inspiratory muscle training
- control group (Sham Comparator): not conduct inspiratory muscle training for 8 weeks
  Interventions: Other: Control group

INTERVENTIONS:
Device: Threshold inspiratory muscle training — Threshold inspiratory muscle training device (Threshold Inspiration Muscle Trainer, Respironics Inc; Pittsburgh, Pennsylvania, USA). The intensiy of IMT was adjusted and verification using Pm measurement in laboratory. Patients spontaneously breathed using resistive-IMT and their Pm were measured simultaneously. Adjusted the intensity of resistive-IMT from small to large according to the Pm waveform. Adjustment completed while mean Pm achieved 60% of MIP and maintained at least 15 minute. Likewise, eligible patients in these group used the resistive IMT device for 15 minutes, twice per day, with an inspiratory load at 60% of PImax as previously adjustment. Training loads were adjusted to maintain 60% of the PImax every week.
  Arms: threshold-IMT group
Device: Resistive inspiratory muscle training — Resistive inspiratory muscle training device(PFLEX, Respironics Inc; Pittsburgh, Pennsylvania, USA). The intensiy of IMT was adjusted and verification using Pm measurement in laboratory. Patients spontaneously breathed using resistive-IMT and their Pm were measured simultaneously. Adjusted the intensity of resistive-IMT from small to large according to the Pm waveform. Adjustment completed while mean Pm achieved 60% of MIP and maintained at least 15 minute. Likewise, eligible patients in these group used the resistive IMT device for 15 minutes, twice per day, with an inspiratory load at 60% of PImax as previously adjustment. Training loads were adjusted to maintain 60% of the PImax every week.
  Arms: resisive-IMT group
Other: Control group — Conventional therapy without any inspiratory muscle training program
  Arms: control group

SUMMARY:
Comparable RCTs of clinical therapeutic effects using respiratory physiology-oriented IMT device in different operation principle in COPD are so far lacking. Therefore the investigators perform an adequately powered RCT on the effects of two IMT device application as an pulmonary physical therapy in patients with COPD with inspiratory muscle weakness.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is defined as sustained expiratory flow limitation small airway disease which is a major cause of morbidity and mortality worldwide. Dyspnoea is the most vital symptom lead to exercise-limiting of COPD which is the major reason of physical activities reduction and consequently contribute to dysfunction of skeletal muscle including diaphragm. Diaphragm sarcopenia is well documented as an important extrapulmonary manifestation of COPD. It has been suggested that reductions in exercise capacity are conversely related to the muscle weakness present in these patients and consequently impact negatively on quality of life. It also contributes to hypoxaemia and hypercapnia in progressive stage.

Mutiple pulmonary rehabilitation programs are regular physical care for stable patients with COPD to improve extrapulmonary disease manifestations. Inspiratory muscle training (IMT) serve as one of pulmonary rehabilitation program that aim at diaphragmatic improvement has been used constantly and is extensively studied in recent years in stable patients with COPD.

From meta-analyses of randomised controlled trials (RCTs) in patients with COPD, it can been concluded that IMT as a stand-alone therapy was proved to increase inspiratory muscle strength and endurance, decrease dyspnea, improve exercise capacity and the quality of life. It was also concluded that COPD patients with inspiratory muscle weakness which defined as PI,max< 60 cmH2O were more likely to significantly improve inspiratory muscle strength and functional exercise capacity when IMT was applied.

IMT is defined as persistent breathing training using the inspiratory training device. Inspiratory muscle trainers were classified into inspiratory resistive trainers® and inspiratory threshold trainers® according to operation principle. The former contain build-in spring-loaded valve which provides a continuous, pre-determined inspiratory load during the entire inspiratory phase; The latter do not provide a constant inspiratory load to ensure the intensity of inspiratory training. There are great differences in operation principle between the two inspiratory muscle trainers above. Inspiratory resistance that generated by inspiratory resistive trainers depend on inspiratory flow rate, however threshold load is independent of inspiratory flow. Intensity of loads in the two IMT devices can be repectively adjust.

However, therapic effect of IMT remains undefined due to disunity of IMT devices and loads in previous studies. Various devices and loads arouses different training intensity which is the key point of securing training effect. The optimized IMT program with proper devices and loads should be figure out. The investigators' previous study elaborated the detailed respiratory physiological response to IMT in COPD. Comparable RCTs of clinical therapeutic effects using respiratory physiology-oriented IMT device in different operation principle in COPD are so far lacking. Therefore the investigators perform an adequately powered RCT on the effects of two IMT device application as an pulmonary physical therapy in patients with COPD with inspiratory muscle weakness.

ELIGIBILITY:
Inclusion Criteria:

1. Severe and very severe COPD (postbronchodilator FEV1/FVC under 70% and FEV1 under 50% of the predicted value (GOLD C and D group);
2. Inspiratory muscle weakness（Maximal Inspiratory Pressure under 60cmH2O）;
3. Bronchial dilation test (BDT) negative;
4. No history of pulmonary rehabilitation.

Exclusion Criteria:

1. severe orthopaedic problems having a major impact on daily activities;
2. previous inclusion in rehabilitation programme (<1 year);
3. diagnosed psychiatric or cognitive disorders
4. progressive neurological or neuromuscular disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle force | 8 weeks
  Maximal inspiratory pressure measurement is a test of inspiratory muscle force. The measurement of maximal inspiratory pressure reflects the strength generated by the entire inspiratory muscles. Patients were normally seated and strongly urged to make maximum inspiratory efforts at residual volume(RV). The maximum pressure value of mouthpiece was measured during the maximal inspiratory maneuvers. The maximum value of three satisfactory manipulation that vary by less than 20% was recorded. Unit of maximal inspiratory pressure measurement is cmH2O (centimeter water column) as a pressure unit.

SECONDARY OUTCOMES:
Health-related quality of life | 8 weeks
  The Chronic Respiratory Disease Questionnaire (CRQ) will be used to assess Health-related Quality of Life(HRQL). This 20-item interviewer-administered questionnaire, which takes about 20 minutes to complete, has a total score and four domain scores (dyspnea, fatigue, emotion, and mastery-the sense of control over the disease). Each item score is 1-7 points, and total score is 20-140 points.
degree of dyspnea | 8 weeks
  The BDI (baseline dyspnea index) and TDI (transition dyspnea index) are interviewer-administered questionnaires that assess dyspnea through its effect on daily activities. The instrument takes about 3 to 4 minutes to complete. The BDI has three scales: functional impairment, magnitude of task, and magnitude of effort. Each is scored on a 0 (severe) to 4 (no impairment) scale. The total score, which sums the three, can therefore range from zero (most limitation from dyspnea) to 12 (no limitation from dyspnea). Changes in limitation in the areas of functional impairment, magnitude of task, and magnitude of effort are rated with the TDI. Each is scored on a -3(major deterioration) to 0(no change) to +3(major improvement) scale.The focal TDI score,which sums the three, therefore, can range from -9(greatest increase in limitation owing to dyspnea)to +9 (greatest reduction in limitation owing to dyspnea).
blood gas analysis | 8 weeks
  Carbon dioxide partial pressure（millimeters of mercury，mmHg） and oxygen saturation（%） were detected and analyzed.
Maximal exercise capacity (incremental cardiopulmonary exercise testing) | 8 weeks
  The maximal incremental exercise tests were conducted on an electrically braked cycle ergometer (Ergoselect 200 K; Cosmed, Rome, Italy) . Symptom-limited-cycle exercise test consisted of a steady-state resting period of 3 min followed by 1 min of unloaded pedaling at 60 cycles/min; the exercise load was increased by 10 Watt each minute, end up while symptom-limited appear. Maximal exercise capacity indexes were analyzed after recording, mainly including the following: endurance exercise capacity(second, s); maximum work(Wmax [Watt, W]) , maximum oxygen uptake (V'O2,max [liter per minute, L/min]), maximum oxygen uptake per kilogram (V'O2,max [milliliters per minute per kilogram, mL/min/kg]), maximal minute ventilation (V'E,max [milliliters per minute, L/min]), carbon dioxide equivalent (V'E/VCO2 [equivalent]).

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Prof, Study Chair — Guangzhou Institute of Respiratory Disease

IPD SHARING:
Plan to Share IPD: Yes